CLINICAL TRIAL: NCT02960451
Title: Randomized Trial of Usual Care vs. Specialized, Phase-specific Care for Youth at Risk for Psychosis
Brief Title: PRIME vs Usual Care for Clinical High Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1411014943
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Clinical High Risk Syndrome for Psychosis
Keywords: prodrome; cognitive behavioral therapy; family focused therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRIME care (Experimental): Specialized care in the PRIME clinic
  Interventions: Other: PRIME care
- Usual care (Active Comparator): Usual care in the community
  Interventions: Other: Usual care

INTERVENTIONS:
Other: PRIME care — Specialist medication, cognitive behavior therapy, family-focused therapy
  Arms: PRIME care
Other: Usual care — Medication and psychotherapy as available form community providers
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether specialty care is superior to usual care in the treatment of patients at clinical high risk for psychosis.

DETAILED DESCRIPTION:
This study is a randomized clinical effectiveness trial for patients at clinical high risk for psychosis that compares two treatments: 1) specialty care delivered in a specialized clinical for patients at clinical high risk for psychosis versus 2) treatment as usual in the community.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following:

  1. Male or female between 12 and 30 years old.
  2. Understand and sign an informed consent (or assent for minors) document in English.
  3. Meet diagnostic criteria for prodromal syndrome as per COPS criteria.

Exclusion Criteria:

* Subjects must not meet any of the following:

  1. Diagnosis of current or lifetime Axis I psychotic disorder, including mood disorder with psychotic symptoms.
  2. Impaired intellectual functioning (full-scale IQ<70). However, those with an IQ in the 65-69 range will not be excluded if they score >75 on the WRAT Reading.
  3. Past or current history of a clinically significant central nervous system disorder that may contribute to prodromal symptoms or confound their assessment.
  4. Alcohol or substance dependence in the past 6 months.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Functioning | 24 months

SECONDARY OUTCOMES:
Service utilization | 24 months
  hospitalizations and emergency room use

CONTACTS AND LOCATIONS:
Overall Officials: Scott Woods, MD, Principal Investigator — Yale University
Locations (1):
- Prevention through Risk Identification Management and Education (PRIME) Clinic, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No